CLINICAL TRIAL: NCT00048425
Title: Randomized, Multicenter Evaluation of Intravenous Levosimendan Efficacy Versus Placebo in the Short Term Treatment of Decompensated Chronic Heart Failure: the REVIVE II Study.
Brief Title: Evaluation of Intravenous Levosimendan Efficacy in the Short Term Treatment of Decompensated Chronic Heart Failure.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3001069
Record Dates: First submitted 2002-10-31; First posted 2002-11-04 (Estimated); Last update posted 2006-12-15 (Estimated); Status verified 2006-12

CONDITIONS: Heart Failure, Congestive
Keywords: Decompensated chronic heart failure
MeSH Terms: conditions — Heart Failure | interventions — Simendan

INTERVENTIONS:
Drug: Levosimendan

SUMMARY:
The purpose of this study is to evaluate the efficacy of a 24-hour infusion of levosimendan compared with placebo in the treatment of decompensated chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* A written informed consent must be obtained for hospitalized male or female patients over 18 years old of age.
* The eligible patients must be diagnosed with worsening heart failure as evidenced by dyspnea at rest, poor ejection fraction and have been treated with IV diuretics.
* It is allowable for the patients to be treated with IV inotropes and vasodilators.

Exclusion Criteria:

The following criteria would exclude the patient from study:

* invasive cardiac procedure (e.g. cardiac surgery, LVAD, cardioversion, cardiac re-synchronization),
* rhythm disorders (e.g. earlier Torsades de Pointes, increased heart rate),
* severe ventricular outflow obstruction,
* angina,
* hypotension,
* uncorrected hypokalemia,
* CNS (e.g. stroke, TIA),
* respiratory (e.g. COPD, intubated patients, oral,
* intravenous or intramuscular steroids),
* renal insufficiency (e.g. increased serum creatinine, dialysis),
* hepatic impairment (e.g. significant increase in liver enzymes),
* decompensation from active infection and acute bleeding (e.g. severe anemia).
* Female patients of child bearing potential must have a negative pregnancy test and use adequate contraceptive precautions.
* Also excluded is the use of amrinone and milrinone prior to randomization, a history of hypersensitivity to levosimendan or any of the excipients and previous participation in a clinical trial with any experimental treatment within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2002-09; Study Completion 2004-12

PRIMARY OUTCOMES:
A clinical composite classification incorporating a Patient Global Assessment at 6 hours, 24 hours and Day 5, combined with clinical criteria for worsening heart failure through 5 days after the start of the study drug infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Krause, Study Director — Abbott
Locations (166):
- United States (132):
  - Cardiovascular Associates/Office of Clinical Research, Birmingham, Alabama
  - Cardiology, P.C. Research, Birmingham, Alabama
  - University Alabama at Birmingham, Birmingham, Alabama
  - Oracle Research-The Heart Center, Huntsville, Alabama
  - Providence Hospital Heart Failure Clinic, Mobile, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - Sarver Heart Center - University of Arizona Health Science, Tucson, Arizona
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Central Cardiology Medical Center, Bakersfield, California
  - Cardiovascular Medical Group & Research Institute, Beverly Hills, California
  - San Diego Cardiovascular Research, Encinitas, California
  - Apex Cardiology Consultants, Inc., Inglewood, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Los Angeles County/USC Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Merced Heart Associates, Merced, California
  - A.R.I. Clinical Trials, Inc., Redondo Beach, California
  - Sacramento Heart and Vascular Research Center, Sacramento, California
  - UCSD Medical Center, University of California, San Diego, California
  - San Diego Cardiac Center, San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - VA Hospital of San Francisco, San Francisco, California
  - Denver Health Medical Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale University School of Medicine/Heart Failure Center, New Haven, Connecticut
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Christiana Care Health System, Newark, Delaware
  - Washington Hospital Center - Cardiac Surgery Department, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Jacksonville Heart Center PA-Baptist Office, Jacksonville, Florida
  - Jacksonville Heart Center,PA, Jacksonville, Florida
  - Watson Clinic Center for Research, Lakeland, Florida
  - MIMA Century Research Associates, Melbourne, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Miami Research & Education Foundation, Miami, Florida
  - The Ford Research Institute PA/NW Florida Heart Group PA, Pensacola, Florida
  - Victor Howard M.D., P.A. Heart Research Center, Port Charlotte, Florida
  - Heart & Vascular Institute of Florida, St. Petersburg, Florida
  - Florida Cardiovascular Institute, Tampa, Florida
  - Augusta Cardiology Clinic, P.C., Augusta, Georgia
  - Memorial Health University Medical Center Research Center, Savannah, Georgia
  - Northwestern Memorial Hospital/Heart Failure Program, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Elgin Cardiology Associates, Elgin, Illinois
  - Midwest Heart Research Foundation, Lombard, Illinois
  - Heart Care Midwest, Peoria, Illinois
  - Clarian Health - Methodist Research Institute Inc., Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - University Hospital, Iowa City, Iowa City, Iowa
  - Via Christi Research Inc. dba PriVia, Wichita, Kansas
  - Gill Heart Institute/University of Kentucky, Lexington, Kentucky
  - Louisiana Heart Center, Chalmette, Louisiana
  - New Orleans Clinical Trial Management, Inc., Covington, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Cardiac Centers of Louisiana, LLC, Shreveport, Louisiana
  - Medical Research Institute, Slidell, Louisiana
  - University of Maryland Hospital, Baltimore, Maryland
  - John Hopkins Bayview Medical Center, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Medical Center, CACR, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Nisus Research/Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Michigan Heart P.C., Ypsilanti, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - VA Medical Center - Cardiology Department, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - St. Paul Clinic, Saint Paul, Minnesota
  - University Hospitals Clinic, Columbus, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - International Heart Institute Montana Foundation, Missoula, Montana
  - Alegent Health Heart and Vascular Institute, Omaha, Nebraska
  - The Creighton Cardiac Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Heart Failure & Transplantation Program, Newark, New Jersey
  - Heart Hospital of New Mexico - NW Heart Institute, Albuquerque, New Mexico
  - Beth Israel Medical Center NY/Phillips Ambulatory Care Center, New York, New York
  - St. Vincent's Hospital, New York, New York
  - Columbia-Presbyterian Medical Center, New York, New York
  - Jack D. Weiler Hospital/Albert Einstein Hospital, The Bronx, New York
  - Montefiore Medical Center/Cardiology Department, The Bronx, New York
  - University Of North Carolina, Chapel Hill, North Carolina
  - The Lindner Center, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation/Department of Cardiology, Cleveland, Ohio
  - OSU Medical Center-Center Wellness & Prevention, Columbus, Ohio
  - The Toledo Clinic & Outpatient Surgery, Toledo, Ohio
  - Toledo Clinic & Outpatient Surgery/Department of Cardiology, Toledo, Ohio
  - Oklahoma Foundation-Cardiovascular, Oklahoma City, Oklahoma
  - University Health Science Center/Cardio Section, Oklahoma City, Oklahoma
  - Hillsboro Cardiology, PC, Hillsboro, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Providence Portland Medical Center/Heart Failure Clinic, Portland, Oregon
  - Geisinger Health System, Danville, Pennsylvania
  - The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Heart Group, Lancaster, Pennsylvania
  - Hahnemann University Hospital/HF and Transplant Center, Philadelphia, Pennsylvania
  - Universtiy of PA Health System, Philadelphia, Pennsylvania
  - Jefferson Heart Institute, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Buxmont Cardiology Associates, Sellersville, Pennsylvania
  - Cardiology Associates of West Reading, West Reading, Pennsylvania
  - Rhode Island Hospital/University Cardiology, Providence, Rhode Island
  - Baptist Clinical Research Center, Memphis, Tennessee
  - Cardiology Group, P.C., Tullahoma, Tennessee
  - Austin-Cardiovascular Associates, Austin, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Cardiopulmonary Research Science & Technology Institute, Dallas, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston VA Medical Center, Houston, Texas
  - St. Luke's Episcopal Hospital/Texas Heart Institute, Houston, Texas
  - Heart Specialists, Nassau Bay, Texas
  - University of Texas Health Sciences, San Antonio, Texas
  - UTHCT/Center for Clinical Research, Tyler, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Carilion Department of Clinical Research, Roanoke, Virginia
  - DUCCS Research of South Boston, South Boston, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - University of Washington, Seattle, Washington
  - Inland Cardiology Associates, Spokane, Washington
  - Southwest Washington Medical Center, Vancouver, Washington
  - Beloit Clinic, SC, Beloit, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (19):
  - Canberra Hospital/Cardiology Department, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital/Department of Cardiology, Camperdown, New South Wales
  - Concord Hospital - Heart Failure Clinic/Department of Cardiology, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Liverpool Hospital - Cardiology Research, Liverpool, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital - Cardiology Department, St Leonards, New South Wales
  - St. George Hospital/Cardiology Department, Sydney, New South Wales
  - Royal Brisbane Hospital - Cardiology Department, Herston, Queensland
  - The Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre - Cardiac Research Department, Bedford Park, South Australia
  - Queen Elizabeth Hospital/Cardiology Department, Woodville, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital/Cardiac Research Unit, Launceston, Tasmania
  - Box Hill Hospital - Coronary Care Unit, Box Hill, Victoria
  - St. Vincent's Hospital - Cardiology Investigational Unit, Fitzroy, Victoria
  - Karinia House/Geelong Hospital, Geelong, Victoria
  - Level 2, Cardiology Department/Royal Melbourne Hospital, Parkville, Victoria
  - Heart Research Institute/Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - Rockyview Hospital, Heart Health Institute, Calgary, Alberta
  - University of Alberta Hospitals, Edmonton, Alberta
  - Neureka Research, Willet Green Niller Centre, Greater Sudbury, Ontario
  - University of Ottawa Health Institute, Ottawa, Ontario
  - Center Hospital University of Sherbrooke, Sherbrooke, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan
- Israel (8):
  - Barzilai Medical Center, Ashkelon
  - Hillel Yaffe Medical Center, Hadera
  - Wolfson Medical Center, Holon
  - Heart Institute, Hadassah MC, Jerusalem
  - EMMS Nazareth Hospital, Nazareth
  - Kaplan Medical Center, Rehovot
  - Sieff Medical Center, Safed
  - Assaf Harofe Medical Center, Zrifin

REFERENCES:
- [Derived] Packer M, Colucci W, Fisher L, Massie BM, Teerlink JR, Young J, Padley RJ, Thakkar R, Delgado-Herrera L, Salon J, Garratt C, Huang B, Sarapohja T; REVIVE Heart Failure Study Group. Effect of levosimendan on the short-term clinical course of patients with acutely decompensated heart failure. JACC Heart Fail. 2013 Apr;1(2):103-11. doi: 10.1016/j.jchf.2012.12.004. Epub 2013 Apr 1. PMID 24621834